CLINICAL TRIAL: NCT05609734
Title: No Cases of Delayed Intracranial Hemorrhage (d-ICH) Among Patients With Mild Traumatic Brain Injury (mTBI) on Oral Anticoagulation Therapy
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: 20HSN3790 nr2
Record Dates: First submitted 2022-10-14; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Traumatic Intracranial Hemorrhage; Traumatic Brain Injury
Keywords: antithrombotic therapy
MeSH Terms: conditions — Intracranial Hemorrhage, Traumatic; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — CT scans, patient journals and bloodsample results, no bloodsamples were saved for further analysizes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with an delayed traumatic intracranial hemorrhage: A total of 249 control CTs was performed, where the initial CT was normal regarding tICH. In the initial assessments 1 case of d-ICH (0,41%) was found, but after second opinion this case (case 1, Table 1) was regarded as a pictorial artefact (Table 1). Hence, no d-ICH was found.
  Interventions: Other: no intervention, only observational retrospective study
- Patients without an delayed traumatic intracranial hemorrhage: A total of 249 control CTs was performed, where the initial CT was normal regarding tICH. In the initial assessments 1 case of d-ICH (0,41%) was found, but after second opinion this case (case 1, Table 1) was regarded as a pictorial artefact (Table 1). Hence, no d-ICH was found.
  Interventions: Other: no intervention, only observational retrospective study

INTERVENTIONS:
Other: no intervention, only observational retrospective study — no intervention, only observational retrospective study

SUMMARY:
Abstract Purpose Patients with anticoagulation therapy has a higher risk of developing traumatic Intracranial Hemorrhage (tICH). Delayed Intracranial Hemorrhage (d-ICH) is a rarer clinical manifestation; however, the incidence varies from 0-9,6 % in other studies. Some studies have also questioned the clinical relevance of d-ICH, since the mortality and the need of neurosurgical intervention is reported to be very low. The aim of this study is to determine the incidence of d-ICH at Sundsvall Regional Hospital.

Methods A retrospective observational study of patients with mTBI and oral anticoagulation therapy. Data from medical records and radiology registry in Sundsvall hospital for 29 months during 2018-2020 in Sundsvall identified 249 patients with an initial negative CT scan who performed a follow-up CT scan. Outcome measure was incidence of d-ICH.

DETAILED DESCRIPTION:
Method This is a retrospective observational study investing the incidence of d-ICH at Sundsvall Regional Hospital. Data was collected from 2018-01-01 - 2020-05-30, and all data collection followed a predetermined protocol. Data was collected by two persons.

Starting from the hospital's radiology registry, all CT-scan referrals from emergency departments surgical section and acute surgical ward with a possible traumatic brain injury was read. Hereafter patients' journals were used to retrieve mechanism of injury, pre-injury medications, and arrival status.

TBI are typically classified after level of consciousness, internationally often measures in Glasgow Coma Scale (GCS) (3). At Sundsvall Regional Hospital, RLS (Reaction Level Scale) is more commonly used, hence it was used in data collection. However, in most cases patients' mental status was only commented as "unaffected" without any use of neither GCS nor RLS. In statistical analysis, we only recorded RLS where it was in clear print and choose not to translate "unaffected" into RLS 1. RLS 1 and GCS 15 are comparable, and GCS 14 and RLS2 are also comparable. mTBI is classified by Scandinavian Neurotrauma Committee's guidelines as a GCS 14 after head trauma, or GCS 15 after head trauma in combination with loss of consciousness, repeated vomiting, posttraumatic seizures, focal neurological deficits, signs of skull fracture, intracranial shunts, antithrombotic treatment, or antiplatelet treatment in combination with age over 65.

Inclusion criteria was mTBI and pre-injury anticoagulation or SGA therapy. In the initial data collection, all patients with mTBI regardless of antitrombotic therapy status were included for comparison for another study. Exclusion criteria was high energy trauma, age <18 years, concealed journals, spontaneous hemorrhage, RLS ≥3 (Figure 1). Due to the lack of control CT, patients on solely ASA or LMWH was also excluded due to former local clinical guidelines.

High energy trauma was excluded from this study, due to the heterogenous variety of injuries and often multiple organ injuries. High energy trauma was defined as any traffic accident or fall > 3 meters, or other traumas that required acute trauma care at the emergency trauma room.

tICH was subcategorized into subdural hemorrhage (SDH), subarachnoid hemorrhage (SAH), epidural hemorrhage or others. Age and gender were collected as demographic data. Severity of head trauma, treatment with anticoagulation therapy (DOAC/VKA/LMWH/other) and/or antiplatelet therapy (ASA/Clopidogrel/Ticagrelor/other) were noted. Antithrombotic therapy was used as an overall term compromising both anticoagulation and antiplatelet treatment. The predominant SGA used for single therapy in Sweden is Clopidogrel, and no participants in this study had single therapy with Ticagrelor. SGA is therefore synonymous with Clopidogrel in this study.

Unclear formulations, positive findings or uncertain findings in the initial radiology assessment was held to a second opinion by an experienced neuroradiologist. A total of 3 cases (1,2 %) were held to a second opinion assessment (Table 1).

Statistics Statistical analysis was executed using Microsoft Excel® version 2108 for Microsoft Windows®. Demographic data were presented as means and standard deviations (SD), or as counts and percentage where appropriate.

The sample size was set to a period of 29 months from January 2018 to May 2020, by which we estimated by the study supervisors to match comparable studies in the field, thus no power calculation prior to study start was done.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria was mTBI and pre-injury anticoagulation or SGA therapy. In the initial data collection, all patients with mTBI regardless of antitrombotic therapy status were included for comparison for another study.

Exclusion Criteria:

* Exclusion criteria was high energy trauma, age <18 years, concealed journals, spontaneous hemorrhage, RLS ≥3 (Figure 1). Due to the lack of control CT, patients on solely ASA or LMWH was also excluded due to former local clinical guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective observational study investing the incidence of d-ICH at Sundsvall Regional Hospital. Data was collected from 2018-01-01 - 2020-05-30, and all data collection followed a predetermined protocol. Data was collected by two persons.
  Starting from the hospital's radiology registry, all CT-scan referrals from emergency departments surgical section and acute surgical ward with a possible traumatic brain injury was read. Hereafter patients' journals were used to retrieve mechanism of injury, pre-injury medications, and arrival status.
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
delayed traumatic intracranial hemorrhage | 6 hours
  Inclusion criteria was mTBI and pre-injury anticoagulation or SGA therapy. A secondary CT scan was performed 6 hours later, to detect a delayed intracranial hemorrhage.

CONTACTS AND LOCATIONS:
Overall Officials: Yücel Cengiz, Ph.D. M.D., Study Director — Umea University
Locations (1):
- Sundsvall Hospital, Sundsvall, Sweden

IPD SHARING:
Plan to Share IPD: No